CLINICAL TRIAL: NCT00446134
Title: Phase 2 Comparison of Weight-based Doses of Taribavirin Combined With Peginterferon Alfa-2b Versus Ribavirin Combined With Peginterferon Alfa-2b in Therapy-naïve Patients With Chronic Hepatitis C Virus Genotype 1 Infection
Brief Title: Taribavirin Phase 2 Dose Finding Study for the Treatment of Hepatitis C Virus (HCV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNA003142-204
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Hepatitis C
Keywords: Phase 2b Dose-Ranging Study
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — taribavirin; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: Drug (Experimental): Oral taribavirin tablet 20 mg/kg/day (Actual doses were 20-24 mg/kg/day) BID plus weekly subcutaneous injections of peginterferon alfa-2b (1.5 ug/kg/wk)
  Interventions: Drug: Taribavirin
- Group 2: Drug (Experimental): Oral taribavirin tablet 25 mg/kg/day (Actual doses were 25-29 mg/kg/day) BID plus weekly subcutaneous injections of peginterferon alfa-2b (1.5 ug/kg/wk)
  Interventions: Drug: Taribavirin
- Group 3: Drug (Experimental): Oral taribavirin 30 mg/kg/day (Actual doses were 30-34 mg/kg/day) BID plus weekly subcutaneous injections of peginterferon alfa-2b (1.5 ug/kg/wk)
  Interventions: Drug: Taribavirin
- Group 4: Drug (Active Comparator): Oral ribavirin 800 mg/day (body weight <65 kg), 1000 mg/day (body weight 65-84 kg), 1200 mg/day (body weight 85-104 kg) or 1400 mg/day (body weight greater than or equal to 105 kg) BID plus weekly subcutaneous injections of peginterferon alfa-2b (1.5 ug/kg/wk)
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Taribavirin — Oral (200 mg) Tablet: 20mg/kg/day BID, patients will be treated for a total of 48 weeks. in addition, all patients will receive peginterferon alfa-2b (PEG-Intron) by weekly subcutaneous injection. Patients who complete treatment with study drug or discontinue treatment prematurely will enter a 24-week follow-up period.
  Other Names: Viramidine; RNA003142-204
  Arms: Group 1: Drug
Drug: Taribavirin — Oral (200 mg) Tablet: 25mg/kg/day BID, patients will be treated for a total of 48 weeks. in addition, all patients will receive peginterferon alfa-2b (PEG-Intron) by weekly subcutaneous injection. Patients who complete treatment with study drug or discontinue treatment prematurely will enter a 24-week follow-up period.
  Other Names: Viramidine; RNA003142-204
  Arms: Group 2: Drug
Drug: Taribavirin — Oral (200mg)Tablet: 30mg/kg/day BID, patients will be treated for a total of 48 weeks. in addition, all patients will receive peginterferon alfa-2b (PEG-Intron) by weekly subcutaneous injection. Patients who complete treatment with study drug or discontinue treatment prematurely will enter a 24-week follow-up period.
  Other Names: Viramidine; RNA003142-204
  Arms: Group 3: Drug
Drug: Ribavirin — Oral (200mg)Tablet: 800 mg/day, 1000 mg/day, 1200 mg/day, or 1400 mg/day BID, patients will be treated for a total of 48 weeks. in addition, all patients will receive peginterferon alfa-2b (PEG-Intron) by weekly subcutaneous injection. Patients who complete treatment with study drug or discontinue treatment prematurely will enter a 24-week follow-up period.
  Other Names: Rebetol; Copegus; Ribasphere; Virazole
  Arms: Group 4: Drug

SUMMARY:
The objective of the study is to select an optimal dose of taribavirin by comparing the efficacy and safety of 3 taribavirin dose levels, 20, 25, and 30 mg/kg/day, versus ribavirin 800 to 1400 mg/day based on body weight, both administered in combination with peginterferon alfa-2b to therapy-naive patients with chronic Hepatitis C Virus (HCV) genotype 1 infection.

DETAILED DESCRIPTION:
The objective of the study is to select an optimal dose of taribavirin by comparing the efficacy and safety of 3 taribavirin dose levels, 20, 25, and 30 mg/kg/day, versus ribavirin 800 mg/day to 1400 mg/day based on subject body weight, with both drugs administered in combination with peginterferon alfa-2b to therapy-naive patients with chronic Hepatitis C Virus genotype 1 infection.

ELIGIBILITY:
Subject Inclusion Criteria

To be eligible for enrollment, patients must meet all of the following criteria:

1. At least 18 years of age
2. Diagnosed with compensated chronic HCV genotype 1 infection that has not been treated with interferon, peginterferon, ribavirin or any experimental therapy for >28 days

2a Serum HCV RNA >2000 copies/mL (780 IU/mL) 2b Liver biopsy performed within 3 years prior to screening consistent with chronic HCV infection 2c Criteria for compensated HCV infection, including normal prothrombin time, serum albumin and bilirubin levels (unless due to non-hepatitis factors) and no history or evidence of bleeding esophageal varices, ascites, or hepatic encephalopathy

3 History of alanine aminotransferase (ALT) elevation either within 6 months prior to screening, at screening, or on retest 2 weeks after a negative screening test, or histologic evidence of HCV infection and a detectable viral load

4 Platelet count ≥90,000/mm3

5 Absolute neutrophil count ≥1200/mm3

6 Hemoglobin ≥12.0 g/dL for females or ≥13.0 g/dL for males

7 Antinuclear antibody (ANA) titer ≤1:320

8 Serum creatinine <1.5 mg/dL

9 HbA1c ≤8.5% for diabetic patients

10 Normal or adequately controlled TSH on prescription medication

11 Alpha fetoprotein (AFP) <20 ng/mL or hepatocellular carcinoma ruled out (ultrasound, CT or MRI scan) within 6 months prior to the study (Patients with an AFP >20 ng/mL must have ongoing hepatocellular carcinoma screening during study as part of the patient's routine medical care)

12 All other clinical laboratory values within normal limits, unless judged not clinically significant by the investigator

13 Sterile or infertile (defined as vasectomy, tubal ligation, postmenopausal, or hysterectomy), or willing to use an approved method of double-barrier contraception (hormonal plus barrier or barrier plus barrier, eg, diaphragm plus condom) from the time of first dose administration until 6 months after the last dose

14 Capable of understanding instructions, adhering to study schedules and requirements, and willing to provided informed consent

Subject Exclusion Criteria

Patients who have any of the following during the screening or Day 1 visit are not eligible for enrollment in this study:

1. Positive HIV or HbsAg serology
2. Severe psychiatric or neuropsychiatric disorders including severe depression, history of suicidal ideations or suicide attempt(s). (This would include patients with a history of suicidal ideations or suicide attempt(s) that occurred when the patient was a minor or many years ago; if the event occurred while under the influence of alcohol or drugs; if the suicidal ideations or suicide attempt(s) were connected to a traumatic event; if the patient was not hospitalized or treated; if the patient has obtained psychiatric clearance for treatment)
3. History or clinical manifestations of significant metabolic, hematological, pulmonary, ischemic or unstable heart disease, gastrointestinal, neurological, renal, urological, endocrine, ophthalmologic (including severe retinopathy), or immune mediated disease
4. History of thalassemia or other hemoglobinopathies (even if the hemoglobin is normal)
5. Chronic hepatic disease other than hepatitis C
6. Organ or bone marrow transplant
7. Chronic (greater than 30 days) use of immunosuppressive medications including steroids in doses equivalent to 10 mg of prednisone or higher, 30 days prior to and anytime during the course of the study
8. Female patients who are breast-feeding or have a positive pregnancy test at any time during the study
9. Males whose female partners are pregnant
10. Patients who have had a malignancy diagnosed and/or treated within the past 5 years, except for localized squamous or basal cell cancers treated by local excision
11. Patients who have participated in a clinical trial and have received an investigational drug within 30 days prior to screening
12. History of alcoholism or drug addiction 1 year prior to screening
13. The use of methadone, buprenorphine or any similar drug, regardless of the prescribed indication or the length of time the patient has been on the drug
14. Chronic (>4 weeks duration) diarrhea, including irritable bowel disease
15. Fibrosis score F4 (cirrhosis) based on Metavir or equivalent index
16. Weight >128 kg or <40 kg
17. Patients infected with mixed HCV genotypes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Poordad, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, 8635 W. 3rd Street, Suite 590W, Los Angeles, California, United States

REFERENCES:
- [Result] Poordad F, Lawitz E, Pozza R, et al. Efficacy and safety of weight-based regimens of taribavirin or ribavirin, given with peginterferon alfa-2b, 12 weeks after treatment (SVR12) in naive patients with genotype 1 hepatitis C. J Hepatol. 2009;50 Suppl 1:S8
- [Result] Poordad F, Lawitz E, Shiffman ML, Hassanein T, Muir AJ, Bacon BR, Heise J, Halliman D, Chun E, Hammond J. Virologic response rates of weight-based taribavirin versus ribavirin in treatment-naive patients with genotype 1 chronic hepatitis C. Hepatology. 2010 Oct;52(4):1208-15. doi: 10.1002/hep.23827. PMID 20721883

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who met all entry criteria and signed an informed consent were randomized in a 1:1:1:1 ratio to one of the 4 arms by a central randomization schedule. A total of 51 clinical centers in the United States participated in the study. 278 patients were randomized; 275 patients who receive one dose of study drug were included in all analyses.
Pre-assignment Details: Randomization was stratified by screening HCV RNA viral load less than or = to 2 or greater than (>) 2 million copies/mL and body weight (BW) (less than or = 75 or >75 kg). A cap of 70% was set for patients with BWs >75 kg so that at least 30% of the patients in each group have BWs less than or = to 75 kg.
Groups:
- Taribavirin 20 mg/kg/Day: Oral taribavirin 20 mg/kg/day (actual doses were 20-24 mg/kg/day) BID plus weekly subcutaneous injections of peginterferon alfa-2b (1.5 ug/kg/wk)
- Taribavirin 25 mg/kg/Day: Oral taribavirin tablet 25 mg/kg/day actual doses were 25-29 mg/kg/day) BID plus weekly subcutaneous injections of peginterferon alfa-2b (1.5 ug/kg/wk)
- Taribavirin 30 mg/kg/Day: Oral taribavirin 30 mg/kg/day actual doses were 30-34 mg/kg/day) BID plus weekly subcutaneous injections of peginterferon alfa-2b (1.5 ug/kg/wk)
- Ribavirin 800 mg/Day: Oral ribavirin 800 mg/day (body weight <65 kg), 1000 mg/day (body weight 65-84 kg), 1200 mg/day (body weight 85-104 kg) or 1400 mg/day (body weight greater than or equal to 105 kg) BID plus weekly subcutaneous injections of peginterferon alfa-2b (1.5 ug/kg/wk)
Period: Overall Study
Arm/Group | Taribavirin 20 mg/kg/Day | Taribavirin 25 mg/kg/Day | Taribavirin 30 mg/kg/Day | Ribavirin 800 mg/Day
Started | 69 (Includes 2 patients who did not receive study drug and was not included in any other analysis) | 70 | 69 (Includes 1 patient who did not receive study drug and was not included in any other analysis) | 70
Completed | 35 | 25 | 26 | 25
Not Completed | 34 | 45 | 43 | 45
Not completed — Adverse Event | 7 | 17 | 13 | 18
Not completed — Lack of Efficacy | 19 | 19 | 24 | 19
Not completed — Protocol Violation | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 3 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 2
Not completed — Adverse Event-Diarrhea | 1 | 1 | 2 | 0
Not completed — Reason Not Completed | 3 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Taribavirin 20 mg/kg/Day | Taribavirin 25 mg/kg/Day | Taribavirin 30 mg/kg/Day | Ribavirin 800 mg/Day | Total
Number analyzed (Participants) | 67 | 70 | 68 | 70 | 275
Age Continuous [Mean (Standard Deviation); unit: years] | 48.5 (9.39) | 47.5 (9.42) | 49.6 (7.24) | 49.7 (8.30) | 48.8 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 25 | 25 | 22 | 107
  Male | 32 | 45 | 43 | 48 | 168
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 4 | 3 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 14 | 13 | 12 | 49
  White | 50 | 41 | 42 | 45 | 178
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 11 | 10 | 11 | 37
Weight [Mean (Standard Deviation); unit: kilograms] | 81.5 (16.9) | 82.6 (16.8) | 82.2 (18.0) | 82.3 (17.1) | 82.1 (17.09)
Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) (log 10) [Mean (Standard Deviation); unit: Copies/mL] | 6.6 (0.71) | 6.6 (0.78) | 6.6 (0.78) | 6.5 (0.84) | 6.6 (0.77)

OUTCOME MEASURES:

1. Primary Outcome: Patients With Either Undetectable Serum HCV RNA (<100 Copies/ml) or at Least a 2-log Decrease From Baseline in Serum Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Treatment Week 12.
Description: The primary efficacy endpoint was the numbers of responders at Treatment Week (TW) 12. Responders are defined as patients achieving either viral negativity or a partial response (PR). Viral negativity is defined as <100 copies/mL serum HCV RNA. A PR is defined as < 100 copies/mL serum HCV RNA and at least a 2-log decrease from baseline in serum HCV RNA levels. Responder rates with corresponding 95% confidence intervals were estimated for each treatment group.
Time Frame: Treatment Week 12
Population: The primary efficacy analysis was performed using the Intent-to-Treat (ITT) population and 275 patients who received at least one dose of study drug were analyzed for efficacy.
Measure: Number; unit: Participants
Arm/Group | Taribavirin 20 mg/kg/Day | Taribavirin 25 mg/kg/Day | Taribavirin 30 mg/kg/Day | Ribavirin 800 mg/Day
Number analyzed (Participants) | 67 | 70 | 68 | 70
Participants
  Early Virologic Response (EVR) (less than 100) | 43 | 40 | 37 | 36
  No EVR (non-responder, Total) | 24 | 30 | 31 | 34
  Detectable (greater than 100 copies/mL at TW 12) | 17 | 17 | 21 | 19
  Discontinued (Prior to TW 12) | 7 | 12 | 10 | 15
  Missing (No value at TW 12) | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Taribavirin 20 mg/kg/Day vs Ribavirin 800 mg/Day; Test type: Non-Inferiority or Equivalence — The study will have 70% to detect non-inferiority of taribavirin versus ribavirin using a non-inferiority margin of 12%; p = 0.167, Fisher Exact; Other = 12.75, 95% CI 2-sided [-3.65 to 29.15], Standard Deviation 5
Statistical Analysis 2: Comparison: Taribavirin 25 mg/kg/Day vs Ribavirin 800 mg/Day; Test type: Non-Inferiority or Equivalence — The study will have 70% to detect non-inferiority of taribavirin versus ribavirin using a non-inferiority margin of 12%; p = 0.611, Fisher Exact; Difference of Proportion = 5.71, 95% CI 2-sided [-10.76 to 22.19], Standard Deviation 5
Statistical Analysis 3: Comparison: Taribavirin 30 mg/kg/Day vs Ribavirin 800 mg/Day; Test type: Non-Inferiority or Equivalence — The study will have 70% to detect non-inferiority of taribavirin versus ribavirin using a non-inferiority margin of 12%; p = 0.736, Fisher Exact; Difference of Proportion = 2.98, 95% CI 2-sided [-13.67 to 19.63], Standard Deviation 5
Statistical Analysis 4: Comparison: Taribavirin 20 mg/kg/Day vs Taribavirin 25 mg/kg/Day; Test type: Non-Inferiority or Equivalence — The study will have 70% to detect non-inferiority of taribavirin versus taribavirin using a non-inferiority margin of 12%; p = 0.485, Fisher Exact; Difference of Proportion = 7.04, 95% CI 2-sided [-9.28 to 23.35], Standard Deviation 5
Statistical Analysis 5: Comparison: Taribavirin 20 mg/kg/Day vs Taribavirin 30 mg/kg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 4]; p = 0.295, Fisher Exact; Difference of Proportion = 9.77, 95% CI 2-sided [-6.72 to 26.26], Standard Deviation 5
Statistical Analysis 6: Comparison: Taribavirin 25 mg/kg/Day vs Taribavirin 30 mg/kg/Day; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 4]; p = 0.864, Fisher Exact; Difference of Proportion = 2.73, 95% CI 2-sided [-13.84 to 19.3], Standard Deviation 5

2. Secondary Outcome: Patients With Anemia (Hemoglobin <10 g/dL) Up to Follow-up Week 24
Description: The primary safety endpoint will be the numbers of patients with hemoglobin <10 g/dL (anemia) at any time during the treatment period. The comparison of anemia rates between taribavirin and ribavirin groups will be carried out using the Fisher's exact test or Chi-square test. The 95% confidence interval of the difference in proportion will be analyzed.
Time Frame: Treatment Week Follow-Up 24
Population: The secondary analysis was performed using the Safety Population and 275 patients who received at least one dose of study drug were analyzed for safety.
Measure: Number; unit: Participants
Arm/Group | Taribavirin 20 mg/kg/Day | Taribavirin 25 mg/kg/Day | Taribavirin 30 mg/kg/Day | Ribavirin 800 mg/Day
Number analyzed (Participants) | 67 | 70 | 68 | 70
Participants | 11 | 11 | 19 | 23
Statistical Analysis 1: Comparison: Taribavirin 20 mg/kg/Day vs Ribavirin 800 mg/Day; Test type: Superiority or Other; p = 0.0304, Chi-squared; Mean Difference (Final Values) = 16.4, 95% CI 2-sided [2.31 to 30.57], Standard Deviation 5
Statistical Analysis 2: Comparison: Taribavirin 25 mg/kg/Day vs Ribavirin 800 mg/Day; Test type: Superiority or Other; p = 0.0293, Chi-squared; Mean Difference (Final Values) = 17.1, 95% CI 2-sided [3.22 to 31.06], Standard Deviation 5
Statistical Analysis 3: Comparison: Taribavirin 30 mg/kg/Day vs Ribavirin 800 mg/Day; Test type: Superiority or Other; p = 0.5816, Chi-squared; Mean Difference (Final Values) = 4.9, 95% CI 2-sided [-10.41 to 20.24], Standard Deviation 5

3. Secondary Outcome: Patients With Undetected Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) (<100 Copies/mL) at Treatment Week Follow-Up 24
Time Frame: Treatment Week Follow-Up 24
Population: This analysis was performed using the Intent-to-Treat Population (ITT); undetectable HCV RNA defined as <100 copies/mL;Patients with a missing value at TW 12, TW 24 were considered Non-responders (detectable); a responder is defined as a patient with undetectable HCV RNA at FW 24 after achieving EVR at TW 12 and undetectable status at TW 24
Measure: Number; unit: Participants
Arm/Group | Taribavirin 20 mg/kg/Day | Taribavirin 25 mg/kg/Day | Taribavirin 30 mg/kg/Day | Ribavirin 800 mg/Day
Number analyzed (Participants) | 67 | 70 | 68 | 70
Participants
  Responder Follow-Up Week 24 | 19 | 19 | 19 | 19
  Non-Responder Follow-Up Week 24 | 48 | 51 | 49 | 51
  Detectable HCV RNA Follow-Up Week 24 | 14 | 15 | 16 | 14
  Discontinued Week Follow-Up Week 24 | 34 | 36 | 33 | 37
Statistical Analysis 1: Comparison: Taribavirin 20 mg/kg/Day vs Ribavirin 800 mg/Day; Test type: Superiority or Other; p = 0.9999, Fisher Exact; Mean Difference (Final Values) = 1.22, 95% CI 2-sided [-13.78 to 16.22], Standard Deviation 5
Statistical Analysis 2: Comparison: Taribavirin 25 mg/kg/Day vs Ribavirin 800 mg/Day; Test type: Superiority or Other; p = 0.9999, Fisher Exact; Mean Difference (Final Values) = 0, 95% CI 2-sided [-14.73 to 14.73], Standard Deviation 5
Statistical Analysis 3: Comparison: Taribavirin 30 mg/kg/Day vs Ribavirin 800 mg/Day; Test type: Superiority or Other; p = 0.9999, Fisher Exact; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-14.11 to 15.71], Standard Deviation 5
Statistical Analysis 4: Comparison: Taribavirin 20 mg/kg/Day vs Taribavirin 25 mg/kg/Day; Test type: Superiority or Other; p = 0.9999, Fisher Exact; Mean Difference (Final Values) = 1.22, 95% CI 2-sided [-13.78 to 16.22], Standard Deviation 5
Statistical Analysis 5: Comparison: Taribavirin 20 mg/kg/Day vs Taribavirin 30 mg/kg/Day; Test type: Superiority or Other; p = 0.9999, Fisher Exact; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-14.76 to 15.59], Standard Deviation 5
Statistical Analysis 6: Comparison: Taribavirin 25 mg/kg/Day vs Taribavirin 30 mg/kg/Day; Test type: Superiority or Other; p = 0.9999, Fisher Exact; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-15.71 to 14.11], Standard Deviation 5

4. Secondary Outcome: Relapsers at Follow-Up Visit 24
Description: Includes patients who had undetectable Hepatitis Virus C (HVC) Ribonucleic Acid (RNA) at their last visit on drug.
Time Frame: Follow-Up Week 24
Population: The analysis was performed using patients who had undetectable HVC RNA at their last visit on drug.
Measure: Number; unit: Participants
Arm/Group | Taribavirin 20 mg/kg/Day | Taribavirin 25 mg/kg/Day | Taribavirin 30 mg/kg/Day | Ribavirin 800 mg/Day
Number analyzed (Participants) | 29 | 24 | 22 | 24
Participants | 10 [-10.08 to 20.86] | 5 [-22.98 to 10.23] | 3 [-28.87 to 17.66] | 5

ADVERSE EVENTS:
Time Frame: Treatment Week Follow-Up 24
Description: A treatment-emergent adverse event (AE) was defined as any AE that began after the first dose of double-blind study study, or began earlier yet worsened after the first dose, to 30 days after the last dose. The AEs were reported by at least 5% of patients in any treatment group and the Safety Population of 275 was used in the analysis.
Arm/Group | Taribavirin 20 mg/kg/Day | Taribavirin 25 mg/kg/Day | Taribavirin 30 mg/kg/Day | Ribavirin 800 mg/Day
Serious Adverse Events (participants affected / at risk) | 7/67 | 6/70 | 6/68 | 9/70
Other Adverse Events (participants affected / at risk) | 66/67 | 68/70 | 68/68 | 69/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taribavirin 20 mg/kg/Day (N=67) | Taribavirin 25 mg/kg/Day (N=70) | Taribavirin 30 mg/kg/Day (N=68) | Ribavirin 800 mg/Day (N=70)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess Jaw (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intentional Self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic Encaphalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Status Epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Distress Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taribavirin 20 mg/kg/Day (N=67) | Taribavirin 25 mg/kg/Day (N=70) | Taribavirin 30 mg/kg/Day (N=68) | Ribavirin 800 mg/Day (N=70)
Fatigue (General disorders) | 44 (44) | 37 (37) | 43 (43) | 36 (36)
Nausea (Gastrointestinal disorders) | 30 (30) | 24 (24) | 29 (29) | 29 (29)
Influenza-like Illness (General disorders) | 20 (20) | 21 (21) | 27 (27) | 24 (24)
Diarrhoea (Gastrointestinal disorders) | 27 (27) | 27 (27) | 25 (25) | 16 (16)
Insomnia (Psychiatric disorders) | 23 (23) | 26 (26) | 23 (23) | 17 (17)
Headache (Nervous system disorders) | 30 (30) | 35 (35) | 22 (22) | 28 (28)
Chills (General disorders) | 17 (17) | 16 (16) | 21 (21) | 14 (14)
Irritability (Psychiatric disorders) | 16 (16) | 12 (12) | 18 (18) | 16 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (21) | 11 (11) | 17 (17) | 14 (14)
Decreased Appetite (Metabolism and nutrition disorders) | 11 (11) | 5 (5) | 17 (17) | 10 (10)
Depression (Psychiatric disorders) | 13 (13) | 24 (24) | 16 (16) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 11 (11) | 15 (15) | 17 (17)
Injection Site Erythema (General disorders) | 20 (20) | 9 (9) | 15 (15) | 17 (17)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 14 (14) | 15 (15) | 23 (23)
Dizziness (Nervous system disorders) | 10 (10) | 18 (18) | 13 (13) | 15 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 11 (11) | 12 (12) | 18 (18)
Pyrexia (General disorders) | 11 (11) | 11 (11) | 12 (12) | 18 (18)
Rash (Skin and subcutaneous tissue disorders) | 11 (11) | 13 (13) | 12 (12) | 12 (12)
Dry Skin (Skin and subcutaneous tissue disorders) | 7 (7) | 14 (14) | 11 (11) | 8 (8)
Neutropenia (Blood and lymphatic system disorders) | 10 (10) | 6 (6) | 11 (11) | 6 (6)
Pain (General disorders) | 6 (6) | 9 (9) | 10 (10) | 8 (8)
Abdominal Pain (Gastrointestinal disorders) | 7 (7) | 10 (10) | 10 (10) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (4) | 9 (9) | 10 (10)
Vomiting (Gastrointestinal disorders) | 11 (11) | 12 (12) | 9 (9) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 10 (10) | 8 (8) | 12 (12)
Pruritis (Skin and subcutaneous tissue disorders) | 11 (11) | 8 (8) | 8 (8) | 13 (13)
Anxiety (Psychiatric disorders) | 8 (8) | 7 (7) | 8 (8) | 7 (7)
Loose Stools (Gastrointestinal disorders) | 7 (7) | 3 (3) | 6 (6) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (8) | 5 (5) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 4 (4) | 5 (5) | 8 (8)
Dysgeusia (Nervous system disorders) | 9 (9) | 4 (4) | 5 (5) | 4 (4)
Injection Site Reaction (General disorders) | 6 (6) | 6 (6) | 3 (3) | 8 (8)
Hypotrichosis (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2) | 3 (3) | 5 (5)
Constipation (Gastrointestinal disorders) | 7 (7) | 6 (6) | 2 (2) | 5 (5)
Sinusitis (Infections and infestations) | 9 (9) | 1 (1) | 1 (1) | 6 (6)
Weight Decreased (Investigations) | 6 (6) | 4 (4) | 5 (5) | 3 (3)
Disturbance in Attention (Nervous system disorders) | 6 (6) | 2 (2) | 6 (6) | 2 (2)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 3 (3) | 2 (2)
Vision Blurred (Eye disorders) | 3 (3) | 5 (5) | 5 (5) | 3 (3)
Asthenia (General disorders) | 5 (5) | 3 (3) | 4 (4) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 4 (4) | 5 (5) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (5) | 1 (1)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 1 (1) | 5 (5)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2) | 1 (1)
Herpes Simplex (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 5 (5) | 1 (1) | 3 (3) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 2 (2) | 3 (3) | 5 (5)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 5 (5)
Injection Site Rash (General disorders) | 1 (1) | 4 (4) | 3 (3) | 0 (0)
Libido Decreased (Psychiatric disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (4) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 1 (1) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 1 (1) | 3 (3)
Memory Impairment (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Mood Swings (Psychiatric disorders) | 2 (2) | 4 (4) | 1 (1) | 3 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 4 (4)
Paraesthesia (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Anger (Psychiatric disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 2 (2)
Injection Site Pruritus (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 5 (5)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Eye Pain (Eye disorders) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Non-cardiac Chest Pain (General disorders) | 1 (1) | 1 (1) | 2 (2) | 6 (6)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 4 (4)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Valeant supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.